CLINICAL TRIAL: NCT01213992
Title: Open-label Pharmacokinetic Study of Iron Isomaltoside 1000 (Monofer®) Administered by 500 mg IV Bolus Injection or 1000 mg Intravenous Infusion to Patients With Non-Dialysis Dependent Chronic Kidney Disease (PK-CKD-03)
Brief Title: Open-label Pharmacokinetic Study of Iron Isomaltoside 1000 (Monofer®) Administered by 500 mg IV Bolus Injection or 1000 mg Intravenous to Patients With CKD
Acronym: PK-CKD-03
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-Monofer-PK-CKD-03; P-Monofer-PK-CKD-03
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Non-dialysis Dependent Chronic Kidney Disease
MeSH Terms: interventions — iron isomaltoside 1000

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monofer® 500 mg (Active Comparator): 500 mg iron isomaltoside 1000
  Interventions: Drug: Iron isomaltoside 1000
- Monofer® 1000 mg (Active Comparator): 1000 mg iron isomaltoside 1000
  Interventions: Drug: Iron isomaltoside 1000

INTERVENTIONS:
Drug: Iron isomaltoside 1000 — Single dose of 500 mg administered as a bolus undiluted over 2 min.
  Arms: Monofer® 500 mg
Drug: Iron isomaltoside 1000 — Single dose of 1000 mg infused over 15 min. The infusion is diluted in 100mL 0,9% sodium chloride
  Arms: Monofer® 1000 mg

SUMMARY:
The purpose of this study is to assess the pharmakokinetic properties of higher doses (500 mg and 1000 mg) of Monofer® in patients suffering from Non-dialysis Dependent Chronic Kidney Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged more than 18 years.
2. Weight above 50 kg.
3. Subjects diagnosed with NDD-CKD with MDRD calculated eGFR between 15-59 mL/min.
4. Hb < 11.0 g/dL.
5. Either or both of the following iron stores indicators below target {Serum ferritin < 100 ug/l and Transferrin saturation (TfS) <20%}.
6. Life expectancy beyond 12 months by Principal Investigator's judgement.
7. Willingness to participate after informed consent.

Exclusion Criteria:

1. Anaemia predominantly caused by factors other than renal impairment or iron deficiency (according to Principal Investigator s' judgment).
2. Iron overload or disturbances in utilization of iron (e.g. haemochromatosis and haemosiderosis).
3. Drug hypersensitivity (i.e. previous hypersensitivity to iron dextran or iron mono- or disaccharide complexes or any excipients of the study drug).
4. Subjects with history of multiple allergies.
5. Decompensated liver cirrhosis and hepatitis (alanine aminotransferase (ALT) > 3 times upper normal limit).
6. History of Immunocompromise and/or history of Hepatitis B and/or C
7. Active acute or chronic infections (assessed by clinical judgment), supplied with white blood cells (WBC) and C-reactive protein (CRP).
8. Rheumatoid arthritis with symptoms or signs of active joint inflammation.
9. Pregnancy and nursing (To avoid pregnancy, women have to be postmenopausal (at least 12 months must have elapsed since last menstruation), surgically sterile, or women of child bearing potential must use one of the following contraceptives during the whole study period and after the study has ended for at least 5 times plasma biological half-life of the investigational medicinal product: Contraceptive pills, intrauterine devices (IUD), contraceptive depot injections (prolonged-release gestagen), subdermal implantation, vaginal ring, and transdermal patches).
10. Extensive active bleeding necessitating blood transfusion.
11. Planned elective surgery during the study.
12. Participation in any other clinical study within 3 months prior to screening.
13. Untreated B12 or folate deficiency.
14. Other I.V. or oral iron treatment or blood transfusion within 4 weeks prior to screening visit.
15. ESA treatment within 8 weeks prior to screening visit.
16. Serum Ferritin > 500 µg/L
17. Any other medical condition that, in the opinion of Principal Investigator, may cause the subject to be unsuitable for the completion of the study or place the subject at potential risk from being in the study or interfere with study drug evaluation. Example, Uncontrolled Hypertension, Unstable Ischemic Heart Disease or Uncontrolled Diabetes Mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Total serum iron pharmakokinetic parameters | 30min, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 24 hours, 48 hours and 72 hours